CLINICAL TRIAL: NCT05690607
Title: Small Volume Blood Testing Validity and Acceptability for HIV-1 and Hepatitis B
Brief Title: Small Volume Blood Testing Validity and Acceptability for HIV-1 and Hepatitis B (TINIES for BBVs)
Acronym: TINIES
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central and North West London NHS Foundation Trust (Other)
Collaborators: British HIV Association (BHIVA) (Unknown)
Responsible Party: Sponsor
Other Study IDs: F-396-2065
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections; Hepatitis B
MeSH Terms: conditions — HIV Infections; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — HBV DNA viral load will be measured from finger prick whole blood collected in microcontainers and compared to standard venepuncture 6ml EDTA tubes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HIV: Phase 1: People (over 18 years) living with HIV-1 attending London Mortimer Market Centre for routine blood tests as part of their HIV care.
  Interventions: Other: Doctors Laboratory TINIES small volume blood testing kit
- HIV: Phase 2: Subset of HIV participants sent TINIES test kit to use in home environment
  Interventions: Other: Doctors Laboratory TINIES small volume blood testing kit
- HBV: Phase 1: People (over 18 years) living with HBV patients attending London Mortimer Market Centre for routine blood tests as part of their HBV care.
  Interventions: Other: Doctors Laboratory TINIES small volume blood testing kit
- HBV: Phase 2: Subset of participants sent TINIES test kit to use in home environment
  Interventions: Other: Doctors Laboratory TINIES small volume blood testing kit

INTERVENTIONS:
Other: Doctors Laboratory TINIES small volume blood testing kit — Doctors Laboratory TINIES small volume blood testing kits comprise microcontainers manufactured by BD Diagnostics designed for sample collection from skin puncture, along with home testing pack with lancets, instructions and Royal Mail postal packs.

SUMMARY:
During the Covid-19 pandemic era, patients indicated that they find a model of care incorporating remote consultations to be acceptable [1-3]. Remote accessibility to care can be enhanced by using new technology to allow small volume testing for routine blood samples. This study aims to prospectively validate the use of small volume blood sampling for routine HIV-1 and Hepatitis B Virus (HBV) viral load (VL), liver function tests (LFTs) and creatinine, and assess the acceptability of this method of blood sampling to people living with HIV (PLWH). These tests form the usual minimum required for safe monitoring on a routine basis to determine viral activity, liver and renal function in patients either on or off antiviral therapy. The UK based Doctors Laboratory TINIES small volume blood testing kits comprise microcontainers manufactured by BD Diagnostics designed for sample collection from skin puncture, along with home testing pack with lancets, instructions and Royal Mail postal packs. We will collect TINIES samples alongside routine venepuncture samples in people attending their routine clinic follow ups. We will then send kits to different participants to collect samples in their own home, along with a follow up questionnaire (written/online). Finally, we will conduct a more in-depth telephone interview for a subset of patients to qualitatively assess acceptability. Routine use of this method of testing could revolutionise care of people living with chronic blood borne viruses, for example HIV and chronic HBV. TINIES could enable remote monitoring, increasing ease of access to care, reducing clinic appointment burden in otherwise healthy individuals, and reduce labour costs in the NHS, for example, by reducing phlebotomy appointments.

DETAILED DESCRIPTION:
Covid-19 has accelerated the move towards increased use of remote healthcare[4]. This model is well-suited to people living with chronic blood borne virus (BBV) infections, as they are often asymptomatic and need only routine monitoring to assess for disease progression, response to treatment and medication adverse effects[5, 6]. However, routine blood tests still require the patient to attend the hospital for venepuncture to collect several 6 millilitre (ml) tubes twice a year. The Covid-19 pandemic led to a decrease in routine blood monitoring for HIV and HBV, due to a combination of the patient and clinician attempting to reduce hospital exposure[2, 7]. This may have a negative impact on patient care due to missed drug toxicity or changes in viral load necessitating drug initiation or changes. Given the post covid-19 shift to remote healthcare for routine appointments is likely to continue in the NHS[1], a mechanism of remote blood monitoring would be beneficial to patients and clinicians.

Screening for syphilis, hepatitis and HIV using home testing with small volume finger prick blood samples has become established in sexual health services [8, 9]. Despite this, home-test finger prick blood sampling use in routine monitoring for patients living with HIV and HBV has not been explored. Finger prick dried blood spots have been investigated as a method of collection for measuring HIV and HBV viral load, particularly in resource-limited settings[10-13]. However, the use of dried blood spots for routine monitoring in high-income setting outpatient clinics is limited by reduced sensitivity in detecting low viral loads, and reduced ability to measure other routine blood tests, including haematology and biochemistry.

There are few published studies investigating HIV-1 viral load measurement on finger prick blood collected in microcontainers, and none investigating HBV viral load. Studies have found self-taken home HIV tests are acceptable to service-users and increase the uptake of HIV testing in key populations, such as MSM and trans people. In contrast, in a London black African community, TINIES for HIV screening were unpopular and it was unfeasible to scale up their use within primary care[16, 17]. Online posting of tests to be self-taken in the home environment is becoming highly acceptable to service users, while recognising this may lead to reduced uptake in certain vulnerable groups[18].

Apart from enabling ongoing monitoring in the event of a future lockdown, there are other reasons why remote testing may be beneficial in clinical care of people living with BBV. Testing at home will reduce the burden of hospital visits for otherwise healthy people, reducing time off work for appointments and travel costs. There may also be a cost reduction for both the UK Health Service (NHS), for example by reducing venepuncture appointments. Stigma of attending the hospital may reduce uptake of regular blood monitoring, and remote testing may overcome this barrier.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 positive patients attending routine clinic follow up at MMC. Patients who are expected to have a detectable viral load will be actively approached.
* Patients with a diagnosis of HBV attending routine outpatient follow up at MMC.
* >18 years of age
* Able to give informed consent

Exclusion Criteria:

* Patients will need to be able to read the instructions, or follow a simple video, for home testing kits

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Majority of people living with HIV (>90%) attending for blood tests will have undetectable viral load, those patients with any of the following criteria will be proactively approached
  * Recent (in last 6 months) HIV VL >50 copies/mL
  * Reporting intermittent (<90% daily) adherence in last 6 months
  * - not currently taking ART
  Conversely, the majority of people living with HBV will have a detectable viral load (due to specific criteria for starting treatment). Therefore, people on treatment for HBV will be proactively approached.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-23 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-01-22 (Estimated)

PRIMARY OUTCOMES:
Detection, sensitivity and specificity of HIV RNA viral load | 6 months
  To determine the limit of detection, sensitivity and specificity of HIV RNA viral load quantification from finger prick whole blood collected in EDTA microcontainers tested when compared to standard venepuncture 6ml EDTA tubes.
Detection, sensitivity and specificity of HBV DNA viral load | 6 months
  To determine the limit of detection, sensitivity and specificity of HBV DNA viral load quantification from finger prick whole blood collected in EDTA microcontainers, compared to standard venepuncture 6ml EDTA tubes.
Feasibility and acceptability of small volume testing for home sampling | 12 months
  To assess the feasibility and acceptability of small volume testing for home sampling for routine blood tests for routine HIV and hepatitis B monitoring.

SECONDARY OUTCOMES:
Assessing concordance between liver function test parameters from finger prick compared to standard venepuncture | 12 months
  Assess concordance between liver function test parameters and creatinine collected from 600µl finger prick compared to standard venepuncture 6ml EDTA tubes
Feasibility for small volume blood samples collected for other experimental markers | 12 months
  Investigate feasibility for small volume blood samples collected for other experimental markers e.g., host response

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Flanagan, MBBS, Principal Investigator — Central and North West London NHS Trust

IPD SHARING:
Plan to Share IPD: Undecided
The study protocol, full study report, anonymised patient level dataset and statistical code for generating the results will be made available to external parties on request.

REFERENCES:
- [Background] Abstracts of the 5th Joint Conference of the British HIV Association (BHIVA) with the British Association for Sexual Health and HIV (BASHH), Virtual, 19-21 April 2021. HIV Med. 2021 Aug;22 Suppl 2:3-126. doi: 10.1111/hiv.13129. No abstract available. PMID 34435437
- [Background] El-Nahal WG, Shen NM, Keruly JC, Jones JL, Fojo AT, Lau B, Manabe YC, Moore RD, Gebo KA, Lesko CR, Chander G. Telemedicine and visit completion among people with HIV during the coronavirus disease 2019 pandemic compared with prepandemic. AIDS. 2022 Mar 1;36(3):355-362. doi: 10.1097/QAD.0000000000003119. PMID 34711737
- [Background] Fung BM, Perumpail M, Patel YA, Tabibian JH. Telemedicine in Hepatology: Current Applications and Future Directions. Liver Transpl. 2022 Feb;28(2):294-303. doi: 10.1002/lt.26293. Epub 2021 Oct 7. PMID 34506686
- [Background] Bestsennyy O, Gilbert G, Harris A, Rost J. Telehealth: A quarter-trillion-dollar post-COVID-19 reality. In: McKinsey Insights. New York: McKinsey & Company; 2021
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] Angus B, Brook G, Awosusi F, Barker G, Boffito M, Das S, et al. BHIVA guidelines for the routine monitoring of adult HIV-1 positive individuals (2019 interim update). In. Herfordshire, UK: British HIV Association; 2019
- [Background] Campbell C, Wang T, Smith DA, Freeman O, Noble T, Varnai KA, Harris S, Salih H, Roadknight G, Little S, Glampson B, Mercuri L, Papadimitriou D, Jones CR, Taylor V, Chaudhry A, Phan H, Borca F, Olza J, Warricker F, Romao L, Ramlakhan D, English L, Klenerman P, Andersson MI, Collier J, Nastouli E, Khakoo SI, Gelson W, Cooke GS, Woods K, Davies J, Barnes E, Matthews PC. Impact of the COVID-19 pandemic on routine surveillance for adults with chronic hepatitis B virus (HBV) infection in the UK. Wellcome Open Res. 2023 Nov 15;7:51. doi: 10.12688/wellcomeopenres.17522.2. eCollection 2022. PMID 38721280
- [Background] Lange B, Roberts T, Cohn J, Greenman J, Camp J, Ishizaki A, Messac L, Tuaillon E, van de Perre P, Pichler C, Denkinger CM, Easterbrook P. Diagnostic accuracy of detection and quantification of HBV-DNA and HCV-RNA using dried blood spot (DBS) samples - a systematic review and meta-analysis. BMC Infect Dis. 2017 Nov 1;17(Suppl 1):693. doi: 10.1186/s12879-017-2776-z. PMID 29143616
- [Background] Jackson K, Tekoaua R, Li X, Locarnini S. Real-world application of the Xpert(R) HBV viral load assay on serum and dried blood spots. J Med Virol. 2021 Jun;93(6):3707-3713. doi: 10.1002/jmv.26662. Epub 2020 Nov 22. PMID 33174623
- [Background] Roger S, Lefeuvre C, Grison M, Ducancelle A, Lunel-Fabiani F, Pivert A, Le Guillou-Guillemette H. Evaluation of the Aptima HBV Quant Dx assay for semi-quantitative HBV viral load from dried blood spots. J Clin Virol. 2020 Aug;129:104524. doi: 10.1016/j.jcv.2020.104524. Epub 2020 Jun 27. PMID 32629186
- [Background] Fong Y, Markby J, Andreotti M, Beck I, Bourlet T, Brambilla D, Frenkel L, Lira R, Nelson JAE, Pollakis G, Reigadas S, Richman D, Sawadogo S, Waters L, Yang C, Zeh C, Doherty M, Vojnov L. Diagnostic Accuracy of Dried Plasma Spot Specimens for HIV-1 Viral Load Testing: A Systematic Review and Meta-analysis. J Acquir Immune Defic Syndr. 2022 Mar 1;89(3):261-273. doi: 10.1097/QAI.0000000000002855. PMID 34732684
- [Background] Fidler S, Lewis H, Meyerowitz J, Kuldanek K, Thornhill J, Muir D, Bonnissent A, Timson G, Frater J. A pilot evaluation of whole blood finger-prick sampling for point-of-care HIV viral load measurement: the UNICORN study. Sci Rep. 2017 Oct 20;7(1):13658. doi: 10.1038/s41598-017-13287-2. PMID 29057945
- [Background] Rossetti R, Smith T, Luo W, Taussig J, Valentine-Graves M, Sullivan P, Ingersoll JM, Kraft CS, Ethridge S, Wesolowski L, Delaney KP, Owen SM, Johnson JA, Masciotra S. Performance evaluation of the Aptima HIV-1 RNA Quant assay on the Panther system using the standard and dilution protocols. J Clin Virol. 2020 Aug;129:104479. doi: 10.1016/j.jcv.2020.104479. Epub 2020 Jun 1. PMID 32531665
- [Background] Dodds C, Mugweni E, Phillips G, Park C, Young I, Fakoya I, Wayal S, McDaid L, Sachikonye M, Chwaula J, Flowers P, Burns F. Acceptability of HIV self-sampling kits (TINY vial) among people of black African ethnicity in the UK: a qualitative study. BMC Public Health. 2018 Apr 13;18(1):499. doi: 10.1186/s12889-018-5256-5. PMID 29653536
- [Background] Seguin M, Dodds C, Mugweni E, McDaid L, Flowers P, Wayal S, Zomer E, Weatherburn P, Fakoya I, Hartney T, McDonagh L, Hunter R, Young I, Khan S, Freemantle N, Chwaula J, Sachikonye M, Anderson J, Singh S, Nastouli E, Rait G, Burns F. Self-sampling kits to increase HIV testing among black Africans in the UK: the HAUS mixed-methods study. Health Technol Assess. 2018 Apr;22(22):1-158. doi: 10.3310/hta22220. PMID 29717978